CLINICAL TRIAL: NCT03895268
Title: Prospective In Vitro Diagnostic Clinical Performance Study for an Influenza A+B Point-of-Care Test Kit on Patients Exhibiting Influenza-like Illness
Brief Title: Influenza A+B Test Kit Performance Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sanwa BioTech Limited (Industry)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: PEP02-03
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Influenza Type A; Influenza Type B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The study will use nasopharyngeal swab specimens taken from hospitalized subjects displaying influenza-like illness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: ALiA Analyser — NPS specimens shall be tested with the investigational device
Device: Influenza A+B Test Kit — NPS specimens shall be tested with the investigational device

SUMMARY:
Prospective clinical study on the performance of an Influenza A+B rapid test kit. The main goal is to establish the sensitivity and specificity (i.e. how accurate the test is) when compared to a gold standard.

Option of participating in this clinical study will be presented to patients displaying influenza-like illness. Informed consent will be collected from patients or patient's next of kin/guardian before samples (nasopharyngeal swab) are taken from the patient.

Nasopharyngeal swabs are tested using both the investigational test kit and a predicate fluorescence immunoassay test kit. All samples will be tested using a molecular-based PCR test kit as a confirmatory test.

The results will be analysed statistically and the performance of the Influenza A+B test kit can be evaluated.

DETAILED DESCRIPTION:
Influenza is an acute respiratory infection caused by influenza viruses which circulate in all parts of the world. Influenza viruses are causative agents of highly contagious, acute, viral infections of the respiratory tract. Influenza viruses are immunologically diverse, single-stranded RNA viruses.

There are 3 types of seasonal influenza viruses, types A, B, and C. Influenza A+B and B viruses circulate and cause outbreaks and epidemics. Influenza type C virus is detected much less frequently and usually causes mild infections, thus presents less significant public health implications.

Seasonal influenza has an incubation period of approximately 2 days and is characterized by a sudden onset of fever, cough, headache, muscle and joint pain, severe malaise, sore throat and a runny nose. Most people recover within a week without requiring medical attention but influenza can cause severe illness or death especially in vulnerable populations such as children, pregnant women and elderlies. Seasonal influenza causes public health concerns as it spreads easily, with rapid transmission in crowded areas including schools and nursing homes.

Antiviral drugs for Influenza A and Influenza B are available in some countries and may reduce severe complications and deaths. Ideally these antiviral drugs need to be administered within 48 hours of onset of symptoms and hence rapid diagnosis of influenza in patients displaying influenza-like Illness can reduce the number of severe complications and deaths associated with influenza.

Fluorescent Immunoassay is a biochemical technique used for detecting the binding of the "detection" antibody and the analyte molecule. The advantages of a fluorescent detection system have been known for many years. These include higher sensitivity detection of the analyte, simplified reagents and simpler assay designs. Several breakthroughs have occurred over the past few years that have enabled the implementation of a fluorescent based immunoassay system at the point of care.

A modern fluorescent based immunoassay uses a fluorescent compound, which absorbs light or energy (excitation energy) at a specific wavelength and then emits light or energy at a different wavelength, as the detection reagent. The difference between the wavelength of the excitation light and the emission light is called the Stokes shift. The greater the shift or difference in the wavelength the less interference there will be by having the excitation light detected as part of the emission light. Recently many technical improvements have occurred that has enabled the implementation of a high sensitivity immunoassay system. These include the availability of narrow wavelength low cost light sources, newer more stable fluorophores that have very wide Stokes shifts, stable solid state light detectors and microprocessors to process and analyse the data from each test.

When a fluorescent detection system is linked to a lateral flow assay and matched with a powerful analyser like the ALiA Diagnostic Platform, the result is improved assay performance, the opportunity for walk away testing along with the elimination of misinterpretation often associated with visually-read point-of-care assays.

Influenza A and Influenza B affect all population, any patients of age 18 or above displaying symptoms of respiratory infection will be included as potential participants.

There will be no restriction on the ethnicity of patients but the majority of patients to be recruited are expected to be of Asian origin as the clinical trial is based in Hong Kong. However, it has been proved that Influenza strains do not vary / have minimal variation in human of different ethnicity.

Study Design:

Option for participating in this clinical study will be presented to patients satisfying the patient selection criteria. Informed consent will be collected from patients before samples (nasopharyngeal swab) are taken.

Nasopharyngeal swabs are tested using the investigational products, a predicate fluorescence immunoassay test, and a molecular-based PCR test will be used as the gold standard.

Study Duration:

Considering the seasonal nature of the disease, duration of the study is estimated to be approximately 24 months from inclusion of first subject to the day of final analysis of the last subject's sample.

Study Hypothesis:

When compared to PCR:

The positive percent agreement (sensitivity) for the investigational product when testing for influenza A and influenza B should be at least 85 percent with a lower bound of the 95 percent confidence interval that is greater than or equal to 70 percent.

The negative percent agreement (specificity) for the Investigational Product when testing for influenza A is at least 90 percent with a lower bound of the 95 percent confidence interval that is greater than or equal to 80 percent.

ELIGIBILITY:
Inclusion Criteria:

* Patient is having NPA collected by the hospital as routine testing
* Patient or patient's next of kin/guardian is willing and able to give informed consent for participation in the trial.
* Patients presented with influenza-like illness, i.e. fever and cough, with onset of illness within 7 days of hospital admission
* Male or Female, 18 years of age or above.

Exclusion Criteria:

• Have had influenza-specific treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Influenza A and Influenza B affect all population, any patients of age 18 or above displaying symptoms of respiratory infection will be included as potential participants.
  There will be no restriction on the ethnicity of patients but the majority of patients to be recruited are expected to be of Asian origin as the clinical trial is based in Hong Kong. However, it has been proved that Influenza strains do not vary / have minimal variation in human of different ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
The clinical sensitivity and clinical specificity of the investigational devices | 2 Years
  Establish clinical sensitivity and specificity of investigational devices by comparing with PCR results using fresh and frozen sample

CONTACTS AND LOCATIONS:
Overall Officials: Paul KS Chan, Prof., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided